CLINICAL TRIAL: NCT03216798
Title: Client and Provider Preferences for HIV Care: Implications for Implementing Differentiated Service Delivery in Thailand
Brief Title: Client and Provider Preferences for HIV Care
Status: Completed | Type: Observational
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Responsible Party: Sponsor
Other Study IDs: Client & Provider Preferences
Record Dates: First submitted 2017-06-23; First posted 2017-07-13 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaires survey — The questionnaires will be self-administered and anonymous. Information obtained from the questionnaire will not contain identifiable information of patients, CBO staff or health care workers.

SUMMARY:
This study will investigate preferences for HIV care among participants enrolled in the "Study to evaluate the feasibility of Community-based Test and Treat strategies among men who have sex with men and transgender women to increase the uptake of HIV testing and treatment services in Thailand" through a model involving linked strategies: The study takes place in four provinces at six sites affiliated with the Thai Red Cross AIDS Research Center (TRCARC): Bangkok (RSAT and SWING), Chiang Mai (CAREMAT), Chonburi (SWING and Sisters) and Songkhla (RSAT). These are all community-based drop-in centers, targeting MSM and TGW.

Participants who are enrolled in the study at any of the TRCARC affiliated sites and who were tested HIV-positive will be invited to participate in the current questionnaire study.

DETAILED DESCRIPTION:
This will be a cross-sectional questionnaire study. A self-administered questionnaire will be used to assess their satisfaction with current clinical services, preferences for location, frequency and provider of HIV services, as well as expectations and concerns.

Furthermore, staff working at the different HIV-care to community-based organizations (CBOs) and the health care workers providing HIV services will be invited to participate as well. They will also be asked to complete a self-administered questionnaire to assess knowledge and attitude, preferences for location, frequency and provider of HIV services, as well as expectation and concerns.

All data collected, from patients, as well as from staff, will be anonymous.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the Community Led Test and Treat Study at either RSAT or SWING
* According to the inclusion criteria of the Community Led Test and Treat Study, participants will be at least 18 years of age
* HIV-infected and receiving ART
* Willing to participate in the survey

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men who have Sex with Men or Transgender women who have been tested HIV-positive in the Community Led Test and Treat Study and are receiving ART.
Sampling Method: Probability Sample
Enrollment: 370 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Preferences for differentiated models of service delivery | 6 months
  A self-administered questionnaire was developed to assess preferences for location, frequency and provider for different aspects of HIV care. For HIV-care to community-based organizations staff and health care workers, additional questions regarding attitudes and knowledge regarding differentiated service delivery will be included.

CONTACTS AND LOCATIONS:
Overall Officials: Nittaya Phanuphak, MD, PhD, Principal Investigator — Thai Red Cross AIDS Research Centre (TRCARC)
Locations (1):
- The Thai Red Cross AIDS Research Centre, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided